CLINICAL TRIAL: NCT03779971
Title: Energy Value of Lentils and Chickpeas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Novotny, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS66-Lentil/Chickpea Study
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-03

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Treatments will be color coded, and samples will be labeled only by subject number and date. Investigators and outcomes assessors will not know the treatments nor the color code until after the data analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): The placebo comparator will be a fully controlled diet made from typical American foods and containing no beans or pulses.
  Interventions: Other: Control Diet
- Lentil (Experimental): The lentil arm will consist of a fully controlled diet made from the same foods as the placebo arm and will also contain lentils.
  Interventions: Other: Lentil Containing Diet
- Chickpeas (Experimental): The chickpea arm will consist of a fully controlled diet made from the same foods as the placebo arm and will also contain chickpeas.
  Interventions: Other: Chickpea Containing Diet

INTERVENTIONS:
Other: Control Diet — Participants will consume a diet prepared and provided by the USDA Nutrition Center. The diet will contain no pulses, legumes, or beans.
  Arms: Control
Other: Lentil Containing Diet — Participants will consume a diet prepared and provided by the USDA Nutrition Center. The diet will contain lentils.
  Arms: Lentil
Other: Chickpea Containing Diet — Participants will consume a diet prepared and provided by the USDA Nutrition Center. The diet will contain chickpeas.
  Arms: Chickpeas

SUMMARY:
This study is being conducted to determine the digestibility of and available energy from pulses.

DETAILED DESCRIPTION:
Previous studies have demonstrated that the metabolizable energy (energy available to the body) from tree nuts is less than predicted by the Atwater factors (the standard approach to determining calorie value of a food). The Atwater approach is over 100 years old and is inaccurate for some foods. This study will be conducted to determine the metabolizable energy from two pulses, lentils and chickpeas. The study will be a human nutrition intervention involving consumption of a controlled diet followed by collection of urine and feces.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 19 and 38 kg/m2
* Age 25 to 75 years during intervention

Exclusion Criteria:

* Known (self-reported) allergy or adverse reaction to study foods
* Women who have given birth during the previous 12 months or who are pregnant/lactating or who plan to become pregnant during the study
* History of bariatric surgery or nutrient malabsorption disease (such as celiac disease), Crohn's disease, diabetes, or metabolic disorders that may interfere with the study
* History of certain cancer diagnosis or treatment in the last 3 years
* Smoking or use of tobacco products in the past 6 months
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Use of certain medications or supplements (prescription or over-the-counter) that may interfere with the study objectives, including blood thinning medications
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Energy excreted in feces and urine | Cumulative from day 10-17
  Energy (units of calories) excreted in feces and urine will be determined by bomb calorimetry.
Energy excreted in feces and urine | Cumulative from day 39-46
  Energy (units of calories) excreted in feces and urine will be determined by bomb calorimetry.
Energy excreted in feces and urine | Cumulative from day 57-64
  Energy (units of calories) excreted in feces and urine will be determined by bomb calorimetry.

SECONDARY OUTCOMES:
Nitrogen excreted in feces and urine | Cumulative from day 10-17, day 39-46, day 57-64
  Nitrogen (g) excreted in feces and urine will be measured.
Fat excreted in feces | Cumulative from day 10-17, day 39-46, day 57-64
  Fat (g) excreted in feces will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Mirecki, MS, Study Director — US Department of Agriculture
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No